CLINICAL TRIAL: NCT04225637
Title: Comparison Between Two Activation Protocols of Miniscrew-Supported Maxillary Expander in Adolescents: A Randomized Controlled Clinical Trial
Brief Title: Comparison Between Two Rates of Activation of Miniscrew-Supported Upper Jaw Expander in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Yomna Mohamed Mohamed Yacout, Assistant lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01012019
Record Dates: First submitted 2020-01-05; First posted 2020-01-13 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Palatal Expansion Technique; Malocclusion; Posterior Crossbite; Maxillary Hypoplasia
Keywords: Rapid Palatal Expansion; Slow Palatal Expansion; Miniscrew; Bone-borne Expander
MeSH Terms: conditions — Malocclusion; Retrognathia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Slow maxillary expansion (Experimental): The miniscrew-supported maxillary expander is activated by turning the expansion screw once every other day.
  Interventions: Device: Miniscrew-Supported Maxillary Expander- Slow activation
- Rapid maxillary expansion (Experimental): The miniscrew-supported maxillary expander is activated by turning the expansion screw twice daily.
  Interventions: Device: Miniscrew-Supported Maxillary Expander- Rapid activation

INTERVENTIONS:
Device: Miniscrew-Supported Maxillary Expander- Slow activation — A maxillary expander is supported on 4 palatal miniscrews. The appliance is activated slowly by turning the expansion screw once every other day to correct the transverse maxillary deficiency.
  Arms: Slow maxillary expansion
Device: Miniscrew-Supported Maxillary Expander- Rapid activation — A maxillary expander is supported on 4 palatal miniscrews. The appliance is activated rapidly by turning the expansion screw twice per day to correct the transverse maxillary deficiency.
  Arms: Rapid maxillary expansion

SUMMARY:
Miniscrew-supported maxillary expanders provide advantages over conventional tooth-supported expanders. However, there is no consensus in the literature regarding their activation protocol. The purpose of the clinical trial is to evaluate and compare the effects of slow and rapid activation rates of miniscrew-supported expanders on the skeletal changes, dento-alveolar changes and the pain experience.

DETAILED DESCRIPTION:
Transverse maxillary deficiency is one of the problems that are commonly encountered in the orthodontic practice. Miniscrew-supported maxillary expansion represents a promising modality for the treatment of transverse maxillary deficiency. However, controversies still exist regarding the activation protocol. One of these controversies is whether using a slow activation protocol would be more beneficial to the patients compared to a rapid activation protocol. Another question that consequently ensues is whether such activation protocol would result in less pain compared to the rapid activation protocol.

The null hypothesis of the current study is that there is no difference between slow and rapid activation protocols of miniscrew-supported expander.

ELIGIBILITY:
Inclusion Criteria:

* Permanent dentition.
* Participants indicated for skeletal maxillary expansion due to unilateral or bilateral posterior cross bite or maxillary transverse deficiency
* Good oral hygiene

Exclusion Criteria:

* History of previous orthodontic or orthopedic treatment
* History of maxillary trauma
* Patients with congenital craniofacial malformations
* Patients receiving pharmacological agents or having systemic diseases that might affect the bone metabolism or the pain response

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Transverse skeletal changes from baseline to an average of 5 months after the initial activation, measured using cone beam computed tomography (CBCT) | At baseline and an average of 5 months after the initial activation
  The data from CBCT scans at the different time points will be exported in Digital Imaging and Communications in Medicine (DICOM) format and processed using suitable software. The relevant landmarks will be defined and located by the investigator to measure the transverse skeletal changes in mm from baseline to the end of passive retention of the expansion.
Dento-alveolar inclination changes from baseline to an average of 5 months after the initial activation, measured using CBCT | At baseline and an average of 5 months after the initial activation
  The data from CBCT scans at the different time points will be exported in DICOM format and processed using suitable software. The relevant landmarks will be defined and located by the investigator to measure the changes in dento-alveolar inclination from baseline to the end of passive retention of the expansion.

SECONDARY OUTCOMES:
Pain score on Numeric Rating Scale (NRS) at baseline | Baseline
  Measures pain and how it affects the daily activities on a NRS where each respondent selects a whole number, between 0 and 10, with 0 being the lowest extreme and 10 being the highest extreme.
Pain score on NRS after the first activation of the maxillary expander | On day 1 after the first activation of the maxillary expander
  Measures pain and how it affects the daily activities on a NRS where each respondent selects a whole number, between 0 and 10, with 0 being the lowest extreme and 10 being the highest extreme.
Pain score on NRS after 1 week of activation of the maxillary expander | After 1 week of activation of the maxillary expander
  Measures pain and how it affects the daily activities on a NRS where each respondent selects a whole number, between 0 and 10, with 0 being the lowest extreme and 10 being the highest extreme.
Pain score on NRS after the last activation of the maxillary expander | At the end of active expansion (an estimated average of 2 to 3 weeks in the rapid expansion group, and 7 to 12 weeks in the slow expansion group)
  Measures pain and how it affects the daily activities on a NRS where each respondent selects a whole number, between 0 and 10, with 0 being the lowest extreme and 10 being the highest extreme.

CONTACTS AND LOCATIONS:
Overall Officials: Yomna M Yacout, BDS, MSc, Principal Investigator — Alexandria University; Nadia M El Harouni, BDS,MSc,PhD, Study Chair — Alexandria University; Essam M Abdallah, BDS,MSc,PhD, Study Chair — Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin L, Ahn HW, Kim SJ, Moon SC, Kim SH, Nelson G. Tooth-borne vs bone-borne rapid maxillary expanders in late adolescence. Angle Orthod. 2015 Mar;85(2):253-62. doi: 10.2319/030514-156.1. Epub 2014 Dec 9. PMID 25490552
- [Background] Yilmaz A, Arman-Ozcirpici A, Erken S, Polat-Ozsoy O. Comparison of short-term effects of mini-implant-supported maxillary expansion appliance with two conventional expansion protocols. Eur J Orthod. 2015 Oct;37(5):556-64. doi: 10.1093/ejo/cju094. Epub 2015 Jan 6. PMID 25564504
- [Background] Lagravere MO, Carey J, Heo G, Toogood RW, Major PW. Transverse, vertical, and anteroposterior changes from bone-anchored maxillary expansion vs traditional rapid maxillary expansion: a randomized clinical trial. Am J Orthod Dentofacial Orthop. 2010 Mar;137(3):304.e1-12; discussion 304-5. doi: 10.1016/j.ajodo.2009.09.016. PMID 20197161
- [Background] Algharbi M, Bazargani F, Dimberg L. Do different maxillary expansion appliances influence the outcomes of the treatment? Eur J Orthod. 2018 Jan 23;40(1):97-106. doi: 10.1093/ejo/cjx035. PMID 28486682
- [Background] Carvalho Trojan L, Andres Gonzalez-Torres L, Claudia Moreira Melo A, Barbosa de Las Casas E. Stresses and Strains Analysis Using Different Palatal Expander Appliances in Upper Jaw and Midpalatal Suture. Artif Organs. 2017 Jun;41(6):E41-E51. doi: 10.1111/aor.12817. Epub 2016 Dec 7. PMID 27925236
- [Derived] ElNaghy R, Al-Qawasmi R, Hasanin M. Do patient-reported outcomes of miniscrew-supported maxillary expansion in adolescent patients differ between slow and rapid activation protocol? Evid Based Dent. 2023 Mar;24(1):28-29. doi: 10.1038/s41432-023-00858-8. Epub 2023 Mar 8. PMID 36890253
- See also: Institutional Review Board (IORG0008839/IRB00010556- Faculty of Dentistry - Alexandria University ) — https://ohrp.cit.nih.gov/search/IrbDtl.aspx